CLINICAL TRIAL: NCT01298037
Title: HBRN: Immune Regulation and Costimulation in Natural History of Chronic Hepatitis B
Status: Active, not recruiting | Type: Observational
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Kyong-Mi Chang, Professor, Gastroenterology, University of Pennsylvania
Other Study IDs: DK082864 HBRN Immunology; U01DK082864 (NIH)
Record Dates: First submitted 2011-02-15; First posted 2011-02-17 (Estimated); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Hepatitis B
Keywords: Immunology, Hepatitis B, HBV
MeSH Terms: conditions — Hepatitis B

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This is an ancillary to the NIDDK-sponsored Hepatitis B Research Network (HBRN) Study Cohort Study NCT01263587. This study will examine the balance between immune regulatory and effector responses in hepatitis B-infected participants enrolled in the HBRN study (NCT01263587).

DETAILED DESCRIPTION:
Aim 1: The clinical and virological status of chronic Hepatitis B (HBV) infection is defined by distinct patterns of immune effector and regulatory responses: The investigators propose that one or more immune regulatory are induced during chronic hepatitis B that define the extent of immune tolerance vs. activation with associated disease activity and viremia. Towards this end, the immune effector and regulatory responses relative to serum HBV DNA, alanine aminotransferase (ALT), Hepatitis B e antigen (HBeAg), Hepatitis B surface antigen (HBsAg) and liver histology will be examined in a cross-sectional manner in patients with chronic HBV and control groups.

Aim 2: Clinical hepatitis flares during chronic hepatitis B reflect altered balance between immune regulatory and effector responses.

ELIGIBILITY:
Inclusion Criteria:

• Providing informed consent for this ancillary study.

Exclusion Criteria:

* Children under 18 years of age, participants with anemia
* Hgb<10 or Hct<30, congestive heart failure or chronic lung disease requiring oxygen, active coronary artery disease with unstable angina, sepsis or renal failure, other significant medical conditions, autoimmune disease or immunosuppression.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will be recruited from multi-site clinical centers in the United States and Canada including primary care hospitals and community centers that have enrolled into the HBRN cohort study (NCT01263587).
Sampling Method: Non-Probability Sample
Enrollment: 201 (Actual)
Dates: Start 2011-02-01 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Immune regulatory and activation measures | 240 weeks
  Immune regulatory and effector responses relative to HBV DNA, ALT and clinical outcome. HBV-specific lymphoproliferative, IFN-gamma and IL 10 responses, T cell activation and costimulatory markers (PD1, CTLA4, CD28, CD127), FoxP3+ Treg frequency, and NK frequency and expression of activating/inhibitory receptors and Dendritic cell frequency.

CONTACTS AND LOCATIONS:
Overall Officials: Kyong-Mi Chang, MD, Principal Investigator — University of Pennsylvania
Locations (12):
- United States (11):
  - California Pacific Medical Center, San Francisco, California
  - University of California San Francisco Medical Center, San Francisco, California
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Minnesota, Plymouth, Minnesota
  - Mayo Clinic Rochester, Rochester, Minnesota
  - University of North Carolina, Chapel Hill, North Carolina
  - University of Texas Southwestern, Dallas, Texas
  - Virginia Commonwealth University, Richmond, Virginia
  - Virginia Mason Medical Center, Seattle, Washington
  - Harborview Medical Center, Seattle, Washington
- University of Toronto, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Hepatitis B Research Network study web site — http://www.hepbnet.org/